CLINICAL TRIAL: NCT05464303
Title: Establishment and Validation of a Standardized Definition for Biliary Atresia Associated Cholangitis After Hepatic Portoenterostomy
Brief Title: Definition for Biliary Atresia Associated Cholangitis After Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Weibing Tang, Dr, Nanjing Children's Hospital
Other Study IDs: ERBAAC
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Biliary Atresia; Cholangitis
MeSH Terms: conditions — Biliary Atresia; Cholangitis | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative cholangitis: Patients who had conducted kasai procedure and suffered from postoperative cholangitis after surgery
  Interventions: Drug: Intravenous Antibodies
- None postoperative cholangitis: Patients who had conducted kasai procedure and followed up in a clinic，at which time they didn't present signs of cholangitis

INTERVENTIONS:
Drug: Intravenous Antibodies — Treatment is usually performed with sensitive third-generation cephalosporins, and medication is adjusted according to blood culture results
  Groups: Postoperative cholangitis

SUMMARY:
Cholangitis is the most common postoperative complication of biliary atresia, with a reported incidence of 40-90%, which seriously affects the surgical effect, survival rate and the quality of life and prognosis of patients. Without of direct evidence, the diagnosis of cholangitis sometimes is difficult to make, thus most of them are diagnosed based on the symptoms of children. According to literature reports, different centers and regions have different diagnostic criteria for postoperative cholangitis after hepatic portoenterostomy, which has a great influence on the accuracy of the incidence rate and appropriate treatment of cholangitis, and also brings differences in the analysis of the causes and prognostic factors of cholangitis.

Based on the above reasons, we used the Delphi method，in which worldwidely 48 experts participated in, to establish the diagnostic scoring system for postoperative cholangitis after biliary atresia.

Now we aimed to verify the specificity and sensitivity of the new scoring system through clinical cases, in order to unify and standardize the diagnostic criteria and provide help for the diagnosis and treatment of cholangitis after biliary atresia.

ELIGIBILITY:
Inclusion Criteria:

① Admission time: 2019.01.01-2021.12.31;

② The first diagnosis after discharge was cholangitis

Exclusion Criteria:

① Cholangitis after non-Kasai procedure;

* Postoperative cholangitis of biliary atresia not operated in the unit; ③ Patient has been treated in other hospitals during this episode; ④ The treatment period for cholangitis is not completed or the patient is discharged automatically.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who had been conducted Kasai procedure have different outcomes. The clinical data of these patients who were diagnosed as cholangitis and were followed up in the clinic were collected in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic cholangitis score | Two years
  The values of the two groups' scores were calculated separately

SECONDARY OUTCOMES:
Score estimates for treatment of cholangitis | Two years
  In the cholangitis group, the correlation between evaluation score and treatment was studied

CONTACTS AND LOCATIONS:
Overall Officials: Tang weibing, Dr, Study Chair — Nanjing Children's Hospital
Locations (1):
- NJMU, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided